CLINICAL TRIAL: NCT02540174
Title: Alcohol and Tobacco Consumption in Patients With Head and Neck or Lung Cancer : Interest of Integrating the Addiction Treatment to the Initial Cancer Treatment Program
Brief Title: Alcohol and Tobacco Consumption in Patients With Head and Neck or Lung Cancer : Interest of an Addiction Treatment
Acronym: ALTAKRA-1405
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Centre Régional de Référence en Cancérologie (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ALTAKRA-1405
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Upper Aerodigestive Tract Neoplasms; Lung Cancer
Keywords: alcohol and tobacco consumption; addiction treatment
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Tobacco Use | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): integrated addiction treatment program
  Interventions: Procedure: integrated addiction treatment program
- Arm B (Other): standard of care
  Interventions: Procedure: standard of care

INTERVENTIONS:
Procedure: integrated addiction treatment program — At the inclusion, a 45 min interview for : the completion of questionnaires (Fagerström, AUDIT, CAST, Socrates, M.I.N.I), the collection of socio-professional information, obstacles and incentives to stop the consumption of alcohol and tobacco, the record of alcohol-tobacco consumptions, the measurement of exhaled carbone monoxide rate expressed in particles per million using the CO tester.
  At 3, 6, and 12 months : a 20 min interview to assess the alcohol-tobacco consumption and the obstacles and incentives to stop the consumption.
  The first addiction consultation will be carried out directly in the cancer treatment unit and integrated to the overall cancer treatment program.
  Arms: Arm A
Procedure: standard of care — The following actions will be performed by a nurse or by the study coordinator on site who have been trained in tobaccology and addictology :
  * At the inclusion, a 45 minutes interview for : the completion of questionnaires (Fagerström, AUDIT, CAST, Socrates, M.I.N.I) , the collection of socio-professional information, obstacles and incentives to stop the consumption of alcohol and tobacco, the record of alcohol-tobacco consumptions, the measurement of exhaled carbone monoxide rate expressed in particles per million (ppm) using the CO tester.
  * At 3, 6, and 12 months: a 20 minutes interview to assess the alcohol-tobacco consumption and the obstacles and incentives to stop the consumption
  Arms: Arm B

SUMMARY:
This is a multicenter, interventional, randomized study among patients with a first lung or head & neck cancer who are still active smokers ± alcohol misusers.The study will aim to compare the systematic implementation of an addiction treatment program initiated at hospital and integrated to the initial cancer treatment program (Arm A), versus the as-usual procedure, which consists in recommendations to follow an addiction treatment program (Arm B)

DETAILED DESCRIPTION:
* Study proposal at the first medical consultation for therapeutic management of a first upper aerodigestive tract cancer or lung cancer.
* Selection criteria validation
* Collection of an informed consent
* Randomization :

Arm A: Experimental arm : Addiction consultation to the overall cancer treatment

Arm B: standard of care

The completion of questionnaires , the measurement of exhaled carbone monoxide rate using a CO tester for all patients, and the integrated addiction treatment among patients randomized in Arm A will not interfere with the medical treatment of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first upper aerodigestive tract cancer or a lung cancer
* Initial cancer treatment
* Aged ≥ 18 and ≤65 years
* Living within a radius of 20 km from the CHRU de Lille/Oscar Lambret Center
* Patient with tobacco addiction: regular smoker = at least 7 cigarettes /week or 1 cigarette/day or short-term ex-smoker = regular smoker who has stopped smoking for less than 1 year from the inclusion date
* Performance status (ECOG/WHO) ≤ 2
* Registered with a social security system
* Informed and signed consent collected before initiation of any study procedures

Exclusion Criteria:

* Previous lung cancer or upper aerodigestive tract cancer
* Previous other cancer < 5 years, evoluting or treated at the inclusion (except uterine cervical carcinoma, basal cell or squamous cell skin carcinoma )
* Mesothelioma and esophageal cancer
* Occasional smoker (less than 7 cigarettes/week or less than 1 cigarette/day)
* Long-term ex-smokers who have stopped smoking for more than 1 year from the inclusion date
* Impossibility to comply with the study procedures due to geographic, social or mental reasons
* Patient under guardianship or tutorship
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Difference in the rates of tobacco abstinent patients at 12 months between arms A and B | 1 year
  to be a "tobacco abstinent" patient has to :
  * be a smoker at the inclusion (M0)
  * declare to be weaned at M6
  * not declare a consumption between M6 and M12
  * a CO rate less than 10 ppm measured with a CO test at M6 and M12
  We compare the two arms in term of tobacco abstinent patients rate.

SECONDARY OUTCOMES:
Frequency of alcohol and tobacco consumptions during the study | initial diagnosis, after 3, 6 and 12 months
  We considere the tobacco and alcohol consumption levels at T0, M3, M6, M12 by the consumption statement and the behaviour change towards tobacco and alcohol, thanks to questionnaires study specific.
Percentage of tobacco abstinent patients at 12 months | 1 year
  to be a "tobacco abstinent" patient has to :
  * be a smoker at the inclusion (M0)
  * declare to be weaned at M6
  * not declare a consumption between M6 and M12
  * a CO rate less than 10 ppm measured with a CO test at M6 and M12
  We calculate the percentage of tobacco abstinent patients at 12 months considering every patient in the trial.
Difference in the rates of alcohol and tobacco abstinent patients at 12 months depending on whether or not they have received an addiction treatment | 1 year
  We use a specialized monitoring in addictology (tobacco/alcohol) at 12 months according to the arms. The information of a monitoring in addictology will be obtained by the study specific questionnaire at M3, M6, M12
Median time between inclusion date and the date of death (from any cause) | 1 year
  Time until progression. The time between the date of inclusion and the date of death whatever the cause is.
Median progression-free time | 1 year
  delay between inclusion date and progression date (clinical or radiological)
Percentage of Arm A patients who attended the addiction treatment program after the first systematic consultation | 1 year
  We note for each patient in arm A if they have at least one addictology specialized consultation after the first consultation which is imposed, during the 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Vannimenus, MD, Study Director — CHRU of Lille
Locations (3):
- France (3):
  - Oscar Lambret Center, Lille
  - CHRU of Lille : Albert Calmette Hospital, Lille
  - CHRU of Lille: Huriez Hospital, Lille

IPD SHARING:
Plan to Share IPD: No